CLINICAL TRIAL: NCT03316118
Title: A Comparison of Analgesic Efficacy of Ultrasound-Guided Genicular Nerve Block Versus Saline Injection for Total Knee Replacement: a Prospective, Randomized Controlled Trial
Brief Title: US Guided GNB vs Saline Injection for TKA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low Enrollment
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Antoun Nader, Principle Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STU#:00204116
Record Dates: First submitted 2017-10-05; First posted 2017-10-20 (Actual); Results first posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Postoperative Pain; Total Knee Arthroplasty; Nerve Block
Keywords: anesthesiology; pain; arthroplasty
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Active Comparator): Patient will receive genicular nerve block with bupivacaine
  Interventions: Drug: bupivacaine
- Group 2 (Placebo Comparator): Patient will receive normal saline as the nerve block
  Interventions: Drug: saline

INTERVENTIONS:
Drug: bupivacaine — Group 1 will receive genicular nerve block using bupivacaine
  Other Names: BUPIV
  Arms: Group 1
Drug: saline — Group 2 will receive genicular nerve block using normal saline
  Other Names: SAL
  Arms: Group 2

SUMMARY:
Do ultrasound-guided genicular nerve blocks with 0.5% bupivacaine provide improved knee analgesia for patients recovering from total knee replacement surgery compared to saline injection?

Hypotheses:

The investigators hypothesize that the combination of ultrasound-guided adductor canal block (ACB) and genicular nerve block will achieve lower opioid consumption and therefore lead to decreased systemic side effects and improved overall satisfaction compared to ultrasound-guided saline injection for patients undergoing minimally invasive elective total knee arthroplasty (TKA).

DETAILED DESCRIPTION:
The study medication and protocol will consist of Group 1 (Active) - ultrasound-guided adductor canal blockade with 10 ml of 0.25% bupivacaine and ultrasound-guided genicular nerve blocks with 6 ml of 0.5% bupivacaine, and Group 2 (Control) - ultrasound-guided adductor canal block with 10 ml of 0.25% bupivacaine and ultrasound-guided genicular nerve blocks with 6 ml of normal saline. The surgeon will be blinded to the subjects study arm assignment.

An ultrasound-guided ACB will be performed at the level of the mid-thigh of the leg halfway between the superior anterior iliac spine and the patella. The femoral artery, femoral vein, saphenous nerve will be visualized by ultrasonography and the expansion of the adductor canal will be recorded. Sensory assessment of the saphenous distribution will be performed at 30 minutes. The ultrasound-guided genicular nerve block will be performed at the site of the superior lateral, the superior medial, and the inferior medial genicular nerves. The superior lateral genicular nerve is located at the confluence of the lateral femoral shaft and the lateral femoral condyle (in the anteroposterior plane) and at the midpoint of the femur (in the lateral plane). The superior medial genicular nerve site is located at the confluence of the medial femoral shaft and the medial femoral condyle (in the anteroposterior plane) and at the midpoint of the femur (in the lateral plane). The inferior medial genicular nerve site is located at the confluence of the medial tibial shaft and the tibial flare (in the anteroposterior plane) and the midpoint of the tibia (in the lateral plane). Color Doppler will be used to identify the arterial structures which serve as landmarks for the corresponding nerves. All nerve blocks will be performed by a study team physician.

Postoperative follow-up will be done by study team member blinded to the group allocation. The dosing of oxycodone/hydrocodone-acetaminophen will be as needed with management goal of a Visual Analog Scale (VAS) score of ≤ 4. Patients with pain not managed by oral agents will receive IV medication. Patients will be visited during their hospital stay every six hours until discharge to record pain scores, opioid consumption, and patient satisfaction. In addition, patients will be given a pain diary to record (VAS) pain scores every six hours until hospital discharge.

A study team member will follow up patients by telephone (if discharged prior to) at 48 hours, 72 hours.

ELIGIBILITY:
Inclusion Criteria:

* Participants 40 to 85 years old who are presenting for minimally invasive total knee arthroplasty under spinal anesthesia and are candidates for peripheral nerve blocks.
* Minimally invasive is defined as custom modified instrumentation, a quadriceps sparing arthrotomy that does not extend beyond 1cm proximal to the patella and surgical techniques that focus on soft tissue protection.

Exclusion Criteria:

* Patient refusal
* American Society of Anesthesiologists physical status classification of 4 or higher
* Pre-existing neuropathy in the femoral or sciatic distribution
* Coagulopathy
* Infection at the site
* Chronic opioid use (greater than 3 months)
* Pregnancy
* Medical conditions limiting physical therapy participation
* Any other contra-indication to regional anesthesia

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antoun M Nader, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Bupivacaine Block: Ultrasound-guided adductor canal blockade with 10 ml of 0.25% bupivacaine and ultrasound-guided genicular nerve blocks with 6 ml of 0.5% bupivacaine
- Saline Sham: Ultrasound-guided adductor canal block with 10 ml of 0.25% bupivacaine and ultrasound-guided genicular nerve blocks with 6 ml of normal saline.
Period: Overall Study
Arm/Group | Bupivacaine Block | Saline Sham
Started | 2 | 0
Completed | 2 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study terminated early due to low enrollment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Continuous [Mean (Full Range); unit: Years] | 71.5 [70 to 73] |  | 71.5 [70 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 |  | 2
  Male | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 2 |  | 2
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 |  | 2
Kilograms (kG) weight [Mean (Full Range); unit: Kilograms] | 95.8 [88 to 103.6] |  | 95.8 [88 to 103.6]
Height Inches [Mean (Full Range); unit: Inches] | 66.5 [66 to 67] |  | 66.5 [66 to 67]
Pre Surgical Baseline Pain at Rest [Mean (Full Range); unit: Units on a scale] — Pre surgical pain in knee reported by subject prior to surgery. VAS scale of 0= no pain to 10 worst pain imaginable).
  Units on a scale | 3 [1 to 5] |  | 3 [1 to 5]

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Opioid Consumption During the Hospital Stay
Description: Post-operative opioid consumption measured in morphine milligram equivalents (MME)during the hospital stay up to 36 hours after surgery.
Time Frame: 36 hours after surgery
Population: Only two subjects enrolled both were randomized to group 1.
Measure: Mean (Full Range); unit: Morphine milligram equivalents (MME)
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 2 | 0
Morphine milligram equivalents (MME) | 24.17 [23 to 27.2] |

2. Secondary Outcome: Mean Pain Scores of the Knee at Rest for the First 48 Hours After Surgery
Description: Mean pain scores post operative reported using the VAS (visual analog scale) for knee pain at rest on a scale of 0 (no pain to 10 worst pain imaginable). This will be assessed every 6 hours up to 48 hours with the visual analog scale where 0 equals no pain and 10 represents excruciating pain.
Time Frame: 48 hours after surgery
Population: Study terminated due to low enrollment. No subjects randomized to group 2.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 2 | 0
score on a scale | 3.05 [2.6 to 3.5] |

3. Secondary Outcome: Overall Satisfaction With Pain Control 72 Hours After Surgery
Description: Overall satisfaction with pain control 72 hours after surgery using a visual analog scale where 0 = not satisfied and 10 being extremely satisfied
Time Frame: 72 hours after surgery
Population: Study terminated early due to low enrollment. No subjects were randomized to group 2.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 2 | 0
score on a scale | 7 [6 to 8] |

4. Secondary Outcome: Length of Hospitalization
Description: Length of hospitalization in hours from time to admission to time of discharge.
Time Frame: Admission to discharge from hospital
Population: Study was terminated early due to low enrollment. No subjects were randomized to group 2.
Measure: Mean (Full Range); unit: Elapsed time in hours
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 2 | 0
Elapsed time in hours | 38.29 [30.57 to 46] |

ADVERSE EVENTS:
Time Frame: 72 hours after surgical procedure.
Description: The study was terminated early. No subjects were randomized to group 2.
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 1/2 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=2) | Group 2 (N=0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Nausea during the post operative period to discharge from the hospital

LIMITATIONS AND CAVEATS:
The limitation to the results is that the study was terminated early for low enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-09-12): https://cdn.clinicaltrials.gov/large-docs/18/NCT03316118/Prot_001.pdf
  • Statistical Analysis Plan (2017-09-12): https://cdn.clinicaltrials.gov/large-docs/18/NCT03316118/SAP_003.pdf